CLINICAL TRIAL: NCT06544135
Title: Use of Thermal Imaging Camera to Assess Perfusion Before and After Vascular Intervention
Acronym: TIC
Status: Recruiting | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY20230726
Record Dates: First submitted 2024-05-08; First posted 2024-08-09 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Arterial Disease; Critical Limb Ischemia; Critical Lower Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- FLIR thermal imaging group: Temperature measurements will be taken of the lower limb using the FLIR camera and correlated with other aspects of each patient.
  Interventions: Device: FLIR One Pro LT

INTERVENTIONS:
Device: FLIR One Pro LT — Thermal imaging camera used to measure temperatures of the lower limb.

SUMMARY:
This is a preliminary prospective observational study measuring change in lower extremity temperature in response to revascularization procedure.

The main question this study aims to answer is:

- Are temperature measurements from a forward looking infrared (FLIR) camera of the lower extremity useful in predicting outcome of revascularization procedures?

DETAILED DESCRIPTION:
This is a preliminary prospective observational study measuring change in lower extremity temperature in response to revascularization procedure.

Patients with lower extremity PAD will be seen in office pre-intervention. Consent to participate in the TIC study will be acquired at this point. Patients will be given a physical copy of their consent form at the time consent is obtained. During this initial visit or subsequent pre-procedural office visit, the smartphone-based thermal camera will be utilized to measure the temperature of the lower extremity foot, ankle, and leg at the plantar, dorsal, and lateral distributions. Comorbidities and demographic factors will be documented from medical records at this time as well.

Data will be gathered at a consistent location to minimize impact of room temperature on measurements.

Patients will then undergo scheduled revascularization with the interventionist.

Post-intervention pictures will be taken immediately after revascularization.

Patients will then be seen again by the research team for follow-up thermal camera imaging, 1 week post-intervention, and weekly post intervention for at least 1 month but up to 6 months.

Thermal measurements will be correlated with intra-op imaging and clinical outcomes in data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Lower extremity peripheral artery disease with tissue loss consistent with Rutherford classification V or VI.
* Planned lower extremity endovascular intervention

Exclusion Criteria:

* Non-arterial ulcers
* Pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People between ages 18 and 99 years with lower extremity peripheral artery disease with a planned endovascular intervention.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change in ABI | Up to 90 days before revascularization; Up to 1 year after revascularization
  Ankle brachial index will be taken before and after intervention and correlated with thermal readings from FLIR.

SECONDARY OUTCOMES:
Major amputations | Up to 1 year after revascularization
  Any associated amputations the subject had after revascularization
Major revascularizations post-initial intervention | Up to 1 year after revascularization
  Any revascularization procedures done after the initial revascularization
Mortality | Up to 1 year after revascularization
  Subject deaths during the length of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jun Li, MD, Principal Investigator — University Hospitals
Locations (3):
- United States (3):
  - University Hospitals Ahuja Medical Center, Beachwood, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio

IPD SHARING:
Plan to Share IPD: No